CLINICAL TRIAL: NCT03036774
Title: Quantitative Ultrasound Assessment of Gastric Volume in Diabetic and Non Diabetic Patients Scheduled for a General Anesthesia
Brief Title: Ultrasound Measure of Gastric Volume in Diabetic and Non Diabetic Patients Before General Anesthesia
Acronym: ECHODIABETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014/30; 2015-A01997-47 (Other: ANSM)
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Diabetes
Keywords: Gastric contents; Ultrasound; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic patient (Experimental): Diabetic patients (type 1 or type 2 diabetes) with scheduled surgery . Ultrasonic measurement of antral area
  Interventions: Procedure: Ultrasonic measurement of antral area
- Non diabetic patient (Other): Patients with scheduled surgery without history of diabetes or a current, treated or untreated, diabetic disease.
  Ultrasonic measurement of antral area
  Interventions: Procedure: Ultrasonic measurement of antral area

INTERVENTIONS:
Procedure: Ultrasonic measurement of antral area — Antral area is measured by ultrasound using a curvilinear abdominal probe of 2-5 MHz and a Logiq E (General Electrics) type echograph or equivalent.
  Ultrasound is done before the induction of general anesthesia. Three consecutive measurements of the anteroposterior (AP) and cranio-caudal (CC) diameters are performed.
  Antral area (CSA expressed in mm²) is show by the following formula: CSA = AP × CC × π / 4.
  Antral area will correspond to the average of the three measures.

SUMMARY:
The main objective is to compare the frequency of a " full stomach " in diabetic patients compared with a control population, all the patients having followed the instructions of preoperative fast.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* American Society of Anesthesiologists (ASA) classification 1 to 3
* Needed a general anesthesia for a programmed surgical intervention
* Respect of instructions of the pre-operative fasting;
* Affiliation to the social security;
* Consent form signed

Non inclusion Criteria:

* Pregnant or breastfeeding women
* Patients already operated or to be operated from the upper digestive tract (esophagus, stomach, duodenum)
* Patients treated with a prokinetic treatment and / or a level 3 analgesic

Exclusion criteria

* Unfeasibility to ultrasound measurement of antral area
* Failure to observe fasting instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with full stomach | one day
  The main objective is to compare the frequency of a "full stomach" in the diabetic population compared to a "control" population just before induction of general anesthesia.
  A "full stomach" is defined by an antral area > 340 mm2
  The main objective is to compare the frequency of a "full stomach" in the diabetic population compared to a "control" population just before induction of general anesthesia.
  A "full stomach" is defined by an antral area > 340 mm2

SECONDARY OUTCOMES:
Glycemia | one day
  To assess the relationship between preoperative blood glucose and gastric emptying in the diabetic population
Fast duration | one day
  To compare the impact of the duration of fasting on the gastric residue in both populations of patients (diabetic and non-diabetic)
Glycated hemoglobin | one day
  To assess the relationship between glycated hemoglobin and gastric emptying in the diabetic population
Evaluation of anxiety using a numerical scale (from 0 -no anxiety- to 10 -maximal anxiety-) | one day
  To compare the impact of anxiety on the gastric residue in both populations of patients (diabetic and non-diabetic) in both populations of patients (diabetic and non-diabetic)
Evaluation of anxiety using a numerical scale (from 0 -no pain- to 10 -maximal pain-) | one day
  To compare the impact of pain on the gastric residue in both populations of patients (diabetic and non-diabetic) in both populations of patients (diabetic and non-diabetic)
Intraoperative hypoxemia | one day
  Evaluation of the risk of intraoperative pulmonary inhalation in both populations of patients (diabetic and non-diabetic)

CONTACTS AND LOCATIONS:
Overall Officials: Julien Rousset, MD, Principal Investigator — Hôpital Tenon; Marc Fischler, MD-PhD, Study Chair — Hôpital Foch; Francis Bonnet, MD-PhD, Study Chair — HopitalTenon
Locations (3):
- France (3):
  - Fondation Ophtalmologique Adolphe de Rotschild, Paris
  - AP-HP Hopital Tenon, Paris
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No